CLINICAL TRIAL: NCT06475599
Title: Efficacy of Anlotinib Hydrochloride Capsules Combined With TQB2450 in the Treatment of Endometrial Cancer in a Randomized, Controlled, Open-label, Multicenter Phase III Clinical Trial
Brief Title: Anlotinib Hydrochloride Capsules Combined With TQB2450 in the Treatment of Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-III-13
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib hydrochloride capsules + TQB2450 injection (Experimental): Anlotinib hydrochloride capsule: 12 mg each time, once a day, oral administration before breakfast, continuous oral administration for 2 weeks and stop for 1 week.
  TQB2450 injection: 1200mg/ time, once every 3 weeks, diluted to 250 mL with normal saline, infusion time was 60±10 minute.
  Interventions: Drug: Anlotinib hydrochloride capsule + TQB2450 injection
- Chemotherapy drug (Active Comparator): Based on each patient's condition and previous treatment history, the investigator will select one of the following chemotherapy drugs for treatment.
  Paclitaxel: dose of 175 mg /㎡, Day 1, every 4 weeks (Q4W). Albumin-bound paclitaxel: dose of 125 mg /㎡, Day 1, Day 8, Day 15, every 4 weeks (Q4W).
  Doxorubicin: dose 60mg/m ², Day1, every 3 weeks (Q3W). Doxorubicin liposome: dose 40mg/ m ²,Day 1, every 4 weeks (Q4W).
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsule + TQB2450 injection — Anlotinib hydrochloride capsule is a multi-target tyrosine kinase inhibitor, which targets VEGFR (VEGFR-1, VEGFR-2 and VEGFR-3), PDGFR, FGFR and c-Kit, etc. It can inhibit tumor progression by inhibiting angiogenesis and tumor growth at the same time.
  TQB2450 injection is a humanized monoclonal antibody targeting programmed death ligand 1 (PD-L1) that prevents the binding of PD-L1 to the PD-1 and B7.1 receptors on the T-cell surface, allowing T-cell reactivation and thus enhancing the immune response.
  Arms: Anlotinib hydrochloride capsules + TQB2450 injection
Drug: Chemotherapy drug — Based on each patient's condition and previous treatment history, the investigator will select one of the chemotherapy drugs (including Paclitaxel, Albumin, Doxorubicin and Doxorubicin hydrochloride) for treatment.
  Arms: Chemotherapy drug

SUMMARY:
To demonstrate that anlotinib hydrochloride capsules combined with TQB2450 injection can significantly prolong progression-free survival (PFS) compared with chemotherapy in patients with recurrent or metastatic endometrial cancer that is non- microsatellite instability high (non-MSI-H) or DNA mismatch repair deficient (non-dMMR).

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic advanced endometrial cancer confirmed by histopathology;
* Patients failed to respond to 1-2 lines of platinum-based doublet-based therapy;
* Provide a traceable MMR/MSI status report or provide biological samples for DNA mismatch repair/microsatellite instability (MMR/MSI) status testing with non-MSI-high (non-MSI-H) or non-dMMR；
* Patients who cannot undergo radical surgery/radiotherapy;
* Age: ≥18 years old (when signing the informed consent); Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0-1; The expected survival time is more than 3 months；
* At least one measurable lesion (RECIST 1.1);
* Good function of the major organs；
* Women of childbearing age should agree that they must use a contraceptive method (e.g. Intra-uterine device (IUD), contraceptive pill, or condom) during the study and for 6 months after the study; A negative serum pregnancy test within 7 days before study entry and must be non-lactating；
* Subjects voluntarily joined this study, signed informed consent, and had good compliance；

Exclusion Criteria:

* Previous use of bevacizumab, endostar, anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, regorafenib, fruquintinib and other anti-angiogenic drugs or immunotherapy drugs targeting programmed cell death protein 1 (PD-1), PD-L1 and other related cells；
* Patients received anti-tumor indications of Chinese patent medicine approved by National Medical Products Administration (NMPA) within 2 weeks before the study treatment；
* Pathology suggested carcinosarcoma (malignant mullerian mixed tumor), endometrial leiomyosarcoma or other high-grade sarcoma, or endometrial stromal sarcoma；
* Hormone therapy for endometrial cancer had been received within 1 week before the first dose of trial medication；
* Surgery, chemotherapy, radiation therapy, or other anticancer therapy had been received within 4 weeks before the initiation of study treatment (the washout period was calculated from the end of the last treatment). The half-life of oral targeted drugs was less than 5 drugs；
* Subjects with known central nervous system metastases and/or carcinomatous meningitis; The patients were not asymptomatic or were treated and stable, had no radiographic evidence of new or expanding brain metastases for at least 2 weeks after treatment for brain metastases, and had discontinued steroids or anticonvulsant therapy for at least 14 days before the initiation of study treatment；
* The patient had developed or had concurrent malignant tumors within the past 3 years；
* Multiple factors that affect the oral administration of anlotinib (e.g., inability to swallow, post-gastrointestinal resection, chronic diarrhea, and intestinal obstruction) may affect the oral absorption of anlotinib；
* Uncontrolled pleural, pericardial, or ascites requiring repeated drainage (investigator judgment); Severe bone injury caused by tumor bone metastasis may occur or occur after enrollment；
* Patients whose imaging (CT or MRI) showed that the tumor had invaded the important blood vessels or the investigators judged that the tumor was likely to invade the important blood vessels and cause fatal hemorrhage during the follow-up study；
* Unmitigated toxic effects higher than CTCAE grade 1 due to any previous antineoplastic therapy, excluding alopecia；
* Major surgical treatment, open biopsy, or significant traumatic injury within 28 days before the first dose；
* A wound or fracture that has not healed for a long time；
* Patients with a history of arterial/venous thrombosis/cancer thrombosis within 6 months before the first dose of drug, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism；
* People who have a history of psychotropic drug abuse and cannot abstain from it or have mental disorders；
* Subjects with any severe and/or uncontrolled illness；
* A history of vaccination with live attenuated vaccine within 28 days before the initiation of study treatment or a planned vaccination with live attenuated vaccine during the study；
* Patients with severe allergic disease, history of severe drug allergy, and known allergic to any component of the trial drug prescription;；
* Active autoimmune disease requiring systemic therapy (e.g., disease-modifying agents, corticosteroids, or immunosuppressive agents) had developed within 2 years before the initiation of study treatment；
* Patients who are diagnosed with immunodeficiency or who are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (at a dose of >10mg/ day of prednisone or other equivalent efficacy hormone) and continue to do so within 2 weeks before the first dose; Major surgical treatment or significant traumatic injury within 4 weeks before the first dose in this study；
* Participated in other clinical trials of antineoplastic drugs within 4 weeks before the first dose；
* Subjects with concomitant diseases that seriously endanger the safety of the subjects or interfere with the completion of the study, or those who were considered to be unsuitable for enrollment for other reasons according to the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by independent imaging review committee (IRC) | Up to 36 months after study start
  Progression-free survival (PFS) as assessed by independent imaging review committee (IRC) according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST1.1) criteria.
  Time from subject randomization (first treatment) to first disease progression or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 36 months after study start
  Time from randomization to death from any cause.
Progression-free survival (PFS) assessed by investigators | Up to 36 months after study start
  Time from subject randomization (first treatment) to first disease progression or death from any cause, whichever occurred first, was assessed by the investigator according to RECIST 1.1.
Objective mitigation rate (ORR) | Up to 36 months after study start
  According to RECIST 1.1 criteria, proportion of patients with confirmed tumor volume reduction to pre-specified values and maintained minimum requirements, namely the proportion of patients with complete response (CR) and partial response (PR).
Duration of Response (DOR) | Up to 36 months after study start
  From the time of tumor first evaluated as complete or partial response to the time of first disease progression or death from various causes，if the tumor remission is not confirmed, it can not be used.
Disease control rate (DCR) | Up to 36 months after study start
  According to RECIST 1.1 criteria, proportion of patients with confirmed tumor volume reduction to pre-specified values and maintained minimum requirements, namely the proportion of patients with CR，PR and stable disease (SD).
Incidence and severity of abnormal laboratory values | Up to 36 months after study start
  Incidence and severity of laboratory inspection indicators exceed the normal range
Incidence and severity of adverse event rate Adverse events (AE), serious adverse event (SAE) | Up to 36 months after study start
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs)
Incidence of dose interruptions, dose reductions, and dose discontinuations due to study-drug-related toxicity during the trial | Up to 36 months after study start
  Incidence of dose interruptions, dose reductions, and dose discontinuations due to study-drug-related toxicity during the trial
Immunogenicity of TQB2450 | Before administration (-15 minutes) in cycles 1, 2, 5, and 9, and 90 days after the last dose (±7days), each cycle is 21 days
  Incidence of anti-drug antibodies (ADAs) and neutralizing antibodies (NAbs)
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) | Up to 96 weeks
  Questionnaire: EORTC Quality of Life Questionnaire (QLQ-C30):For questions 1 to 28, choose a number from 1 to 4, 1 means none and 4 means very good. For questions 29 and 30, choose a number from 1 to 7, with 1 being very poor and 7 being very good.
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | Up to 96 weeks
  Questionnaire: European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) : The scale has numbers from 0 to 100. 100 represents the best health imaginable. 0 is the worst health imaginable.
European Organization for Research on Treatment of Cancer Endometrial cancer Specific scale QLQ-EN24 | Up to 96 weeks
  Questionnaire: European Organization for Research on Treatment of Cancer Quality of Life questionnaire 24 (QLQ-EN24)：From questions 1 to 24, choose a number from 1 to 4, where 1 means none and 4 means very much.

CONTACTS AND LOCATIONS:
Locations (61):
- China (61):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Guigang City People's Hospital, Guigang, Guangxi
  - Nanxishan Hospital of Guangxi Zhuang Autonomous Region, Guilin, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Liuzhou Municipal Liutie Central Hospital, Liuchow, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hainan Ceneral Hospital, Haikou, Hainan
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang first People's Hospital National Third Class A Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Central Hospital Of Shaoyang, Shaoyang, Hunan
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - Changchun Tumor Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - General Hospital Of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai Red Cross Hospital, Xining, Qinghai
  - The Second Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Binzhou People's Hospital, Binzhou, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Yidu Central Hospital Of Weifang, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Tengzhou Central People's Hospital, Zaozhuang, Shandong
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Maternal Health School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - The Southwest Hospital of Amu, Chongqing
  - Chongqing University Three Gorges Hospital, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Affiliated Hospital of Southwest Medical University, Chongqing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tianjin Central Hospital of Gynecology Obstetrics, Tianjin